CLINICAL TRIAL: NCT00902902
Title: A Clinical Study of GP73 as a HCC Early Tumor Mark
Brief Title: A Clinical Study of GP73 as a Hepatocellular Carcinoma (HCC) Tumor Mark
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Dr. Yilei Mao, Peking Union Medical College Hospital
Other Study IDs: PUMCH-Liver surgery -GP73
Record Dates: First submitted 2009-05-13; First posted 2009-05-15 (Estimated); Last update posted 2009-05-15 (Estimated); Status verified 2009-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: Hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Human serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- 1
- 2

SUMMARY:
The aims of this study were divided into three parts:

1. To evaluate the sensitivity and specificity of GP73 for the diagnosis of hepatitis B related HCC. Established the standard of GP73 in normal people.
2. To definitude the connections between the GP73 level and various diseases.
3. To find the relations of HCC metastasis and recurrence.

Study design:

1. Collectivity type: Prospective，randomized, controlled, multi-central clinical study.
2. Patients: The subjects were from different hospitals including: Peking Union Medical College Hospital (PUMCH), The Cancer Hospital of Peking Union Medical College (PUMC), QiDong Cancer Institute, and Department of Surgery University of Chicago from November of 2007 till the end of this study.

Study arrangement:

This study was consisted of three parts:

1. Established the standard of normal people and test the sensitivity and specificity of HCC patients. The samples were acquired from Health Screen Center and Department of liver surgery of PUMCH, The Cancer Hospital of PUMC and QiDong Cancer Institute.
2. Extend the study bound, including the hepatitis B virus (HBV) and hepatitis C virus (HCV) carriers. The HBV (+) samples were come from Chinese hospitals and institutions. The HCV (+) samples were provide by the Department of Surgery University of Chicago.
3. Research the relations of serum GP73 level and the other diseases, such as other malignant liver tumors, liver metastatic tumors, liver benign tumor, HCC recurrence following surgery etc.

ELIGIBILITY:
Inclusion Criteria:

* A group of patients with no history of liver disease, alcohol consumption less than 40g a week, and no risk factors for viral hepatitis were enrolled from the General Internal Medicine clinics. All subjects in this control group were documented to have normal liver biochemistry.
* Consecutive patients with HCC and patients with HBV & HCV that were age, gender, and race/ethnicity matched to the HCC patients were enrolled from the Liver Clinic during this period. The diagnosis of HCC was made by histopathology, and if histopathology was not available by two imaging modalities (ultrasound [US], magnetic resonance imaging [MRI], or computed tomography) showing a vascular enhancing mass >2cm. HBV infection status was based on hepatitis B surface antigen (HBsAg). HCV infection status was based on serum HCV antibody and HCV-RNA positive.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The subjects were from different hospitals including: Peking Union Medical College Hospital, The Cancer Hospital of PUMC, QiDong Cancer Institute, and Department of Surgery University of Chicago from November of 2007 till the end of this study.
Sampling Method: Probability Sample
Enrollment: 0 (Estimated)
Dates: Start 2008-01; Primary Completion 2008-12 (Actual); Study Completion 2009-07 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- The University of Chicago, Chicago, Illinois, United States